CLINICAL TRIAL: NCT00302146
Title: Functional Imaging in Subjects With Glucocerebrosidase Mutations
Brief Title: Positron Emission Tomography (PET) Imaging in People With Gaucher Mutations
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060055; 06-HG-0055
Record Dates: First submitted 2006-03-11; First posted 2006-03-13 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-03-18

CONDITIONS: Parkinson Disease; Gaucher Disease
Keywords: Lysosomal Storage Disorder; Carrier; L-Dopa Uptake; Glucocerebrosidase; Pathogenesis; Natural History; Gaucher Disease; Healthy Volunteer; HV
MeSH Terms: conditions — Parkinson Disease; Gaucher Disease; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Asymptomatic: Unaffected at-risk individuals with or without a first degree family member with parkinsonism, GD with and without a family history of PD, Gaucher carriers with and without a family history of PD.
  Interventions: Drug: 15-0 H20
- Control: Controls will include subjects without GBA mutations, with sporadic PD and healthy volunteers who do not have a family history of parkinsonism or Gaucher disease.
  Interventions: Drug: 15-0 H20
- PD: Subjects with parkinsonism to better characterize the parkinsonian phenotype (e.g.,GD/PD, Sporadic PD, Gaucher carrier PD).
  Interventions: Drug: 15-0 H20

INTERVENTIONS:
Drug: 15-0 H20

SUMMARY:
This study will use positron emission tomography (PET) to compare how people with Gaucher disease or Gaucher disease carriers with parkinsonism, and their family members, use dopamine in their brains in comparison with healthy normal volunteers and people who have Parkinson disease. PET assesses organ function by measuring metabolism. In this study, magnetic resonance imaging (MRI) is used in conjunction with PET to help better interpret and understand the information gleaned from PET.

People 21 years of age and older with the following conditions may be eligible for this study:

* Gaucher disease and parkinsonism
* Parkinsonism and a family history of Gaucher disease
* Gaucher disease and a family history of parkinsonism
* Gaucher disease carriers who have parkinsonism or a family history of parkinsonism
* Unaffected people with a family history of Gaucher disease and parkinsonism
* Healthy volunteers

Participants undergo the following tests and procedures:

* Personal and family medical history
* Physical examination
* PET scan: The subject lies on a table that slides into the PET scanner until his or her head is positioned properly in the scanner. A catheter is inserted into a vein. An initial scan is done to obtain images before radionuclides are injected. Radioactive water is then injected through the catheter and the subject is asked questions in order to stimulate blood flow in certain areas of the brain to show what parts of the brain are activated. Fluorodopa is then infused through the catheter over 3 minutes. The PET scan can last up to 2 hours.
* MRI scan: This test uses a magnetic field and radio waves to obtain images of organs. The subject lies still on a bed in the middle of a circular scanner for about 30 minutes.

DETAILED DESCRIPTION:
An association between Gaucher disease and parkinsonism has been demonstrated by the concurrence of parkinsonian manifestations in patients with Gaucher disease and an increased incidence of glucocerebrosidase (GBA1) mutations in subjects with parkinsonism of various ethnicities. Furthermore, there are a significant number of obligate and confirmed Gaucher carriers with parkinsonian manifestations. In 2009, an international collaborative study demonstrated that the odds ratio for carrying a GBA1 mutation in subjects with PD was 5.43 (95% CI, 3.89 to 7.57), confirming definitively that mutations in this gene are a common risk factor for PD. A subsequent study in cohorts with Dementia with Lewy bodies showed that the odds ratio (>8) for carrying a GB1mutation was even higher in this associated synucleinopathy. However, in affected and at-risk individuals, the identification and characterization of early parkinsonian manifestations, and the rate of progression of symptoms have not been studied comprehensively and longitudinally. This in-vivo study employs multiple imaging modalities to better define the phenotype in GBA1-associated parkinsonism, follow disease progression, and identify at-risk individuals. The subjects include patients with Gaucher disease and Gaucher carriers with parkinsonian manifestations. In addition, clinically unaffected but at-risk individuals carrying GBA mutations, with and without a family history of parkinsonism will also be included. The control groups consist of individuals with Gaucher disease but no parkinsonian symptoms and relatives of probands without GBA mutations as well as PD patients without GBA mutations and healthy volunteers enrolled in NIMH clinical protocols. Positron emission tomography (PET) with 6-[F-18] Fluoro-L-Dopa (6FD) is used to evaluate presynaptic dopaminergic function, where 6FD uptake in putamen and striatum is employed as a measure of neuronal structural integrity in the substantia nigra. H(2)^15O PET is used to evaluate changes in resting regional cerebral blood flow (rCBF) associated with regional changes in cortical synaptic activity and metabolism. Each subject is screened with an MRI to rule-out anatomic brain abnormalities, and to further delineate areas of interest in the PET scans. Subjects also undergo transcranial ultrasonography (TCS) to assess the substantia nigra. The results of both the PET scans and TCS will be kept confidential, and will not be communicated to the individuals or families involved in the study. In addition to the imaging studies, all patients will undergo a physical and neurological examination, neurocognitive evaluation, olfactory testing and will be surveyed for potential non- motor manifestations.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study will include adult subjects age 21 or older. There will be two major study groups. The first will include subjects with parkinsonism to better characterize the parkinsonian phenotype and the second group will have unaffected yet at-risk individuals with or without a first degree family member with parkinsonism to explore early signs and symptoms of disease.

Control subjects will include individuals without GBA1 mutations. Subjects with sporadic PD and healthy volunteers who do not have a family history of parkinsonism or Gaucher disease will be enrolled as control subjects.

Healthy volunteers and control subjects with parkinsonism will be matched for age, gender and handedness for statistical purposes. When available, we would like to study unaffected siblings (without GBA1 mutations) of parkinsonian subjects. Sib-pair studies will especially be valuable to exclude both environmental and other genetic risk factors for the development of parkinsonian manifestations.

EXCLUSION CRITERIA:

Subjects excluded from the study include those:

1. with severe cognitive deficits impairing decision making at time of enrollment without an appointed surrogate decision maker.
2. who are unable or it is medically unsafe to withdraw from their current medications, such as subjects on psychoactive medications. The subjects on medications that may affect CNS function may be included in the study only with an approval from the prescribing physician to discontinue their medications temporarily for the study.
3. pregnant or nursing. All women of child bearing potential will undergo a pregnancy test.
4. with a history of neurologic conditions such as stroke or any focal brain lesion that may result in parkinsonian manifestations, including subjects with deep brain stimulators
5. cannot lie on his/her back for a prolonged period of time

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult subjects age 21 or older. There will be two major study groups. The first will include subjects with parkinsonism to better characterize the parkinsonian phenotype and the second group will have unaffected yet at-risk individuals with or without a first degree family member with parkinsonism to explore early signs and symptoms of disease. Control subjects will include individuals without GBA1 mutations. Subjects with sporadic PD and healthy volunteers who do not have a family history of parkinsonism or Gaucher disease will be enrolled as control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2006-05-23 (Actual)

PRIMARY OUTCOMES:
Imaging techniques | Ongoing
  Imaging techniques will evaluate whether there are early changes in cerebral L-Dopa stores associated with glucocerebrosidase mutations in subjects with and without parkinsonism.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Sidransky, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
pending
Supporting Information: Study Protocol
Time Frame: pending
Access Criteria: pending

REFERENCES:
- [Background] Neudorfer O, Giladi N, Elstein D, Abrahamov A, Turezkite T, Aghai E, Reches A, Bembi B, Zimran A. Occurrence of Parkinson's syndrome in type I Gaucher disease. QJM. 1996 Sep;89(9):691-4. doi: 10.1093/qjmed/89.9.691. PMID 8917744
- [Background] Tayebi N, Walker J, Stubblefield B, Orvisky E, LaMarca ME, Wong K, Rosenbaum H, Schiffmann R, Bembi B, Sidransky E. Gaucher disease with parkinsonian manifestations: does glucocerebrosidase deficiency contribute to a vulnerability to parkinsonism? Mol Genet Metab. 2003 Jun;79(2):104-9. doi: 10.1016/s1096-7192(03)00071-4. PMID 12809640
- [Background] Wong K, Sidransky E, Verma A, Mixon T, Sandberg GD, Wakefield LK, Morrison A, Lwin A, Colegial C, Allman JM, Schiffmann R. Neuropathology provides clues to the pathophysiology of Gaucher disease. Mol Genet Metab. 2004 Jul;82(3):192-207. doi: 10.1016/j.ymgme.2004.04.011. PMID 15234332
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-HG-0055.html